CLINICAL TRIAL: NCT01632163
Title: A Randomized, Double-blind, Placebo-controlled, 2-arm Parallel-group, Multicenter Study With a 24-week Treatment Period Assessing the Efficacy and Safety of Lixisenatide in Patients With Type 2 Diabetes Insufficiently Controlled With Basal Insulin With or Without Metformin
Brief Title: Assessment of the Efficacy and Safety of Lixisenatide in Patients With Type 2 Diabetes Insufficiently Controlled With Basal Insulin +/- Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC12382; U1111-1124-1213 (Other: UTN)
Record Dates: First submitted 2012-06-26; First posted 2012-07-02 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Experimental): 24-week treatment with lixisenatide once daily on top of basal insulin with or without metformin (at least 1.0g/day)
  Interventions: Drug: Lixisenatide (AVE0010)
- Placebo (Placebo Comparator): 24-week treatment with placebo once daily on top of basal insulin with or without metformin (at least 1.0g/day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Pharmaceutical form:solution
  Route of administration: subcutaneous injection
  Arms: Lixisenatide
Drug: Placebo — Pharmaceutical form:solution
  Route of administration: subcutaneous injection
  Arms: Placebo

SUMMARY:
Primary Objective:

- To assess the effects on glycemic control of lixisenatide in comparison to placebo as an add-on treatment to basal insulin with or without metformin in terms of HbA1c reduction over a period of 24 weeks in insufficiently controlled type 2 diabetic patients.

Secondary Objectives:

* To assess the effects of lixisenatide over 24 weeks on :

  * percentage of patients reaching HbA1c<7% or ≤6.5%,
  * 2-hour postprandial plasma glucose (PPG) and plasma glucose (PG) excursions during standardized meal challenge test,
  * fasting plasma glucose (FPG),
  * change in 7-point self-monitored plasma glucose (SMPG) profile),
  * body weight,
  * change in daily basal insulin dose.
* To assess lixisenatide safety and tolerability.
* To assess anti-lixisenatide antibody development.

DETAILED DESCRIPTION:
Maximum study duration of approximately 35 weeks ± 9 days (up to 2 weeks screening + 8 weeks run-in + 24 weeks double-blind treatment+ 3 days follow-up)

ELIGIBILITY:
Inclusion criteria :

- Patients with type 2 diabetes mellitus (T2DM) diagnosed for at least 1 year at the time of the screening visit insufficiently controlled with basal insulin± metformin.

Exclusion criteria:

At screening:

* Age < legal age of adulthood.
* HbA1c<7% or >10.5%.
* Basal insulin treatment has not been at a stable regimen for at least 3 months and at a stable dose (± 20%) of at least 15 U/day for at least 2 months prior to screening visit.
* If metformin is given, metformin treatment has not been at a stable dose of at least 1.0 g/day for at least 3 months prior to screening visit.
* History of hypoglycemia unawareness.
* Body Mass Index (BMI) ≤20 kg/m².
* Use of other oral or injectable glucose-lowering agents other than basal insulin or metformin within 3 months prior to the time of screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | from baseline to week 24

SECONDARY OUTCOMES:
Percentage of patients with HbA1c <7%, =<6.5% | at week 24
Change in 2-hour postprandial plasma glucose and plasma glucose excursion | from baseline to week 24
Change in fasting plasma glucose | from baseline to week 24
Change in 7-point self monitoring plasma glucose profile (average and each point) | from baseline to week 24
Change in body weight | from baseline to week 24
Change in daily basal insulin dose | from baseline to week 24
Number of patients with adverse events | 24 weeks
Anti-lixisenatide antibody assessment | from baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (51):
- China (30):
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156033, Beijing
  - Investigational Site Number 156006, Beijing
  - Investigational Site Number 156005, Beijing
  - Investigational Site Number 156004, Beijing
  - Investigational Site Number 156002, Beijing
  - Investigational Site Number 156016, Changchun
  - Investigational Site Number 156025, Changsha
  - Investigational Site Number 156014, Chengdu
  - Investigational Site Number 156013, Chengdu
  - Investigational Site Number 156034, Dalian
  - Investigational Site Number 156035, Fuzhou
  - Investigational Site Number 156021, Guangzhou
  - Investigational Site Number 156023, Haikou
  - Investigational Site Number 156017, Harbin
  - Investigational Site Number 156026, Jinan
  - Investigational Site Number 156029, Jinan
  - Investigational Site Number 156019, Nanjing
  - Investigational Site Number 156020, Nanjing
  - Investigational Site Number 156018, Qingdao
  - Investigational Site Number 156028, Shanghai
  - Investigational Site Number 156007, Shanghai
  - Investigational Site Number 156032, Shenyang
  - Investigational Site Number 156009, Shijiazhuang
  - Investigational Site Number 156036, Siping
  - Investigational Site Number 156010, Suzhou
  - Investigational Site Number 156008, Tianjin
  - Investigational Site Number 156027, Wuhan
  - Investigational Site Number 156011, Xi'an
  - Investigational Site Number 156012, Xi'an
- India (10):
  - Investigational Site Number 356019, Ahmedabad
  - Investigational Site Number 356018, Aligarh
  - Investigational Site Number 356026, Bangalore
  - Investigational Site Number 356017, Bhubaneswar
  - Investigational Site Number 356002, Hyderabad
  - Investigational Site Number 356024, Hyderabad
  - Investigational Site Number 356015, Nagpur
  - Investigational Site Number 356008, Pune
  - Investigational Site Number 356021, Secunderabad
  - Investigational Site Number 356023, Visakhapatnam
- Russia (5):
  - Investigational Site Number 643007, Kirov
  - Investigational Site Number 643003, Saint Petersburg
  - Investigational Site Number 643004, Saint Petersburg
  - Investigational Site Number 643005, Saint Petersburg
  - Investigational Site Number 643006, Samara
- South Korea (6):
  - Investigational Site Number 410003, Daegu
  - Investigational Site Number 410007, Goyang
  - Investigational Site Number 410006, Seoul
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410002, Wŏnju

REFERENCES:
- [Derived] Yao J, Zhang M, Zhang X, Zhang J. Impact of Type 2 Diabetes Duration on the Efficacy and Safety of Add-on Lixisenatide in Asian Individuals Receiving Basal Insulin: A Pooled Analysis. Diabetes Ther. 2023 Apr;14(4):653-669. doi: 10.1007/s13300-023-01369-6. Epub 2023 Feb 21. PMID 36809495
- [Derived] Yang W, Min K, Zhou Z, Li L, Xu X, Zhu D, Venkateshwar Rao A, Murthy LS, Zhang N, Li I, Niemoeller E, Shang S. Efficacy and safety of lixisenatide in a predominantly Asian population with type 2 diabetes insufficiently controlled with basal insulin: The GetGoal-L-C randomized trial. Diabetes Obes Metab. 2018 Feb;20(2):335-343. doi: 10.1111/dom.13072. Epub 2017 Oct 5. PMID 28742225